CLINICAL TRIAL: NCT00805909
Title: A Phase IIa, Open-Label, Dose-Titration, Multicenter Study to Assess the Safety and Preliminary Efficacy of NI-0401 in Patients With Acute Cellular Renal Allograft Rejection
Brief Title: NI-0401 in Patients With Acute Renal Allograft Rejection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Light Chain Bioscience - Novimmune SA (Industry)
Responsible Party: Penny Ward/Study Director, NovImmune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NI-0401-02
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Acute Renal Transplant Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NI-0401 (Experimental): 5 daily infusions of escalating doses of NI-0401
  Interventions: Drug: NI-0401

INTERVENTIONS:
Drug: NI-0401 — 5 daily infusions with escalating doses of NI-0401

SUMMARY:
The purpose of the study is to determine the safety and tolerability of NI-0401 and whether NI-0401 can reverse BpACR.

ELIGIBILITY:
Main inclusion Criteria:

* evidence of cellular rejection in a renal biopsy according to Bannff 97 criteria
* rise in Serum Creatinine concentration by >20% compared to baseline value

Main Exclusion Criteria:

* previous therapy with anti-CD3 mAB(OKT3) or anti-lymphocytes polyclonal antibodies (ATG, Atgam)
* patients with cardiac insufficiency or fluid overload
* severe HLA sensitization (>50% panel reactive antibodies prior transplantation)
* defined concomitant disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Nature,frequency,intensity,causality and seriousness of adverse events | Studay day 1 to week 6

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Necker, Paris, France